CLINICAL TRIAL: NCT07082582
Title: Investigating in Humans the Impact of Training Status on Dietary Consumption With Direct Measurement of Ingestive Behaviour
Acronym: HITS
Status: Recruiting | Type: Observational
Sponsor: Michele Serra (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, Michele Serra, Clinical Research Manager, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: 2024-00926
Record Dates: First submitted 2025-06-17; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Food Intake Regulation; Training Status
Keywords: Ingestive behavior; Gut Hormones; Drinkometer
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples are collected from venous blood before, directly after, and 30 minutes after the meal test. Plasma samples will be isolated from blood samples and stored at -80° C for later analysis. The analysis of DNA is not planned in this study. Nevertheless, plasma can contain cell-free DNA (cfDNA). Considering that no solution for the stabilisation of nucleic acid is added to the plasma samples, a complete or meaningful sequencing of the cfDNA can hardly be expected from the plasma samples collected in this study.
  Stool samples are collected at two different time points to establish the circadian rhythm of the gut microbiome. Metagenomics and metatranscriptomics analysis will be performed only on microbial genetic material.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants with trained Status: Trained status: continuous participation in a structured training program for at least the past six months, in addition to meeting the minimum requirement of physical activity of 150 min of moderate physical activity or 75 min of vigorous physical activity per week.
- Participants with untrained Status: Untrained status: No participation in any structured training program for the last six months, in addition to not performing physical activity above 150 min of moderate physical activity or 75 min of vigorous physical activity per week.

SUMMARY:
The goal of the research project is to investigate the influence of training status on ingestive behavior and postprandial physiological responses in the human body. The investigators aim to understand how regular training influences the choice and amount of food consumed, as well as the associated physiological processes, including changes in the spectrum of gut hormones. The investigators are particularly interested in how these factors differ between individuals who train regularly compared to those who do not follow a structured training program.

The research project aims to translate findings from previous animal experiments to humans and to examine whether and how training affects food handling and physiological responses, similar to observations made in rodents. This information could significantly contribute to improving recommendations for diet and physical activity in the population.

DETAILED DESCRIPTION:
The goal of the proposed research is to identify the differences in ingestive behavior that might be caused by the training status in humans after long-term structured exercise. For this, the investigators plan to investigate and cross-sectionally compare microstructural parameters of ingestive behavior between individuals with trained and untrained status when offered three different meals (high-carbohydrate, high-fat, high-sucrose lactose-free milk) separately or concurrently.

Furthermore, the investigators propose to explore a possible correlation between microstructural parameters of ingestive behavior and postprandial levels of several gut hormones, and to investigate the differences in the composition and activity of the gut microbiome between the two groups, especially in relation to the observed ingestive behavior. Finally, the investigators will investigate the relationship between ingestive behavior and body composition separately for the two groups.

The microstructure of ingestive behavior of both male and female individuals in relation to training status has never been investigated in a direct measurement approach before and the investigators of this project are the only one that currently have both the technical requirements as well as the necessary experience to carry out such studies.

The previous research project "Direct measurement of changes in food selection and intake behavior after RYGB surgery" (NCT04933305, NCT03747445) was successful. Although recruitment and retention of study participants was significantly hindered by the COVID-19 pandemic after March 2020, the investigators were able to publish four peer-reviewed scientific articles out of the proposed studies so far. Four additional manuscripts are currently in preparation.

The present research project builds logically on previous work in the field of bariatric surgery and builds a new collaborations with Prof. J. Nicholas Betley and Dr. Lavinia Boccia (University of Pennsylvania, USA). This collaboration will surely lead to relevant findings which will be published in at least two peer-reviewed publications.

ELIGIBILITY:
Inclusion Criteria:

* Training status classified as "trained" or "untrained",
* Chronological age ≥ 18 and ≤ 35,
* Body Mass Index ≥ 18.5 and ≤ 26,
* Current enrolment in a university,
* Language: English or German, with a sufficient English proficiency to fill out the food questionnaire,
* Ability and willingness to participate in the study, and
* Voluntarily signed informed consent.

Exclusion Criteria:

* History of previous metabolic and bariatric surgery,
* Current use of medications for medical treatment (excluding contraceptive measures),
* Current use of over-the-counter medications for weight loss or appetite control,
* Current medical diagnosis of metabolic disorders (such as type

  1 or 2 diabetes mellitus),
* Use of antibiotics in the last two months,
* History of use of probiotics (excluding yogurt and sauerkraut),
* Smoking,
* Biological or surgical menopause,
* Polycystic ovary syndrome (PCOS),
* Pregnancy, lactation, or current attempt of conception, and
* History of chronic substance abuse.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Participants in the trained group are recruited from a rowing club affiliated with the University of Zürich (UZH) and Federal Technical institute of Zürich (ETH).
  Participants in the untrained group are recruited from students and employees of UZH and ETH.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Energy Intake from Liquid Meal Consumption | From enrolment to the end of the study participation through four study visits within three months.
  Total energy intake (in kilocalories) from consumption of high-carbohydrate, high-sucrose, and high-fat lactose-free milk during each visit. Intake is measured using a drinkometer device that quantifies the exact volume consumed, which is then converted into kilocalories based on the known energy density of each meal type. The unit of measure is kilocalories (kcal).
Macrostructure of Ingestive Behavior (Rate of Energy Intake) | From enrolment to the end of the study participation through three of four study visits within three months
  The rate of energy intake is calculated for each participant during the ingestion of each of the three test stimuli, based on standardized measurements from the drinkometer system. This measure reflects the average caloric intake per second over the course of the test stimulus consumption. Energy intake is determined by the volume of liquid consumed, multiplied by the known caloric density of the test stimulus, and divided by the duration of the ingestion period. The unit of measure is kilocalories per second (kcal/s).
  This outcome is assessed during the first three study visits, in which a single test stimulus is administered at each visit. It is not measured during the fourth study visit, where all three test stimuli are presented simultaneously.
Macrostructure of Ingestive Behavior (Meal Duration) | From enrolment to the end of the study participation through three of four study visits within three months.
  Meal duration is defined as the total time taken by each participant to consume each of the three test stimuli, measured using the standardized drinkometer system. For each stimulus, the duration is recorded from the initiation of ingestion (first measurable suck) to the completion of consumption (last measurable suck). The unit of measure is seconds (s).
  This outcome is assessed during the first three study visits, each involving the administration of a single test stimulus. Meal duration is not measured during the fourth study visit, where all three test stimuli are offered to participants simultaneously.
Macrostructure of Ingestive Behavior (Number of Sucks) | From enrolment to the end of the study participation through three of four study visits within three months.
  The primary outcome is the number of sucks performed by each participant during the ingestion of each of the three test stimuli, as measured using a standardized drinkometer system. A "suck" is defined as a discrete negative pressure event generated by the participant to draw in liquid, as detected by the drinkometer's calibrated weight sensors. For each stimulus, the total number of sucks is recorded as a simple count, with the unit of measure being "number (n)." The outcome is assessed during the first three study visits, each of which features a single test stimulus administered in a standardized fashion. This outcome is not measured during the fourth study visit, in which all three test stimuli are offered simultaneously to the participant.
Microstructure of Ingestive Behavior (Suck Energy Intake) | From enrolment to the end of the study participation through three of four study visits within three months.
  Suck energy intake is defined as the total amount of energy (in kilocalories) consumed by the participant during each individual suck, measured for each of the three test stimuli using a standardized drinkometer system. For each test stimulus, the total caloric intake is calculated by multiplying the volume of liquid ingested by its caloric density and summing the values across all measured sucks. The unit of measure is kilocalories (kcal).
  This outcome is assessed during the first three study visits, where each visit involves a single test stimulus. Suck energy intake is not measured during the fourth study visit, in which all three test stimuli are presented to the participant simultaneously.
Microstructure of Ingestive Behavior (Suck Duration) | From enrolment to the end of the study participation through three of four study visits within three months.
  Suck duration is defined as the time span of each individual suck performed by the participant during the ingestion of each of the three test stimuli, as measured by a standardized drinkometer system. For each test stimulus, the duration of every suck is recorded from the initiation to the completion of the negative pressure event. The unit of measure is seconds (s).
  This outcome is assessed during the first three study visits, where a single test stimulus is administered at each visit. Suck duration is not measured during the fourth study visit, in which all three test stimuli are presented simultaneously.
Microstructure of Ingestive Behavior (Suck Rate) | From enrolment to the end of the study participation through three of four study visits within three months.
  Suck rate is defined as the average energy intake of liquid ingested per second during each individual suck, measured for each of the three test stimuli using a standardized drinkometer system. For each test stimulus, the energy intake consumed during each suck is divided by the corresponding suck duration to determine the rate of ingestion for that event. The unit of measure is kilocalories per second (kcal/s).
  This outcome is assessed during the first three study visits, where a single test stimulus is administered at each visit. Suck rate is not measured during the fourth study visit, in which all three test stimuli are presented simultaneously.
Microstructure of Ingestive Behavior (Suck Maximal Rate) | From enrolment to the end of the study participation through three of four study visits within three months.
  Suck maximal rate is defined as the highest instantaneous rate of liquid ingestion (in kilocalories per second) achieved during any single suck by the participant for each of the three test stimuli, as measured using a standardized drinkometer system. For each test stimulus, the maximal rate is determined by identifying the suck with the greatest energy intake per unit time among all measured sucks during the ingestion period. The unit of measure is kilocalories per second (kcal/s).
  This outcome is assessed during the first three study visits, with each visit involving a single test stimulus. Suck maximal rate is not measured during the fourth study visit, where all three test stimuli are presented simultaneously.
Microstructure of Ingestive Behavior (Burst Number) | From enrolment to the end of the study participation through three of four study visits within three months.
  Burst number is defined as the total count of distinct bursts performed by the participant during the ingestion of each of the three test stimuli, as measured using a standardized drinkometer system. A "burst" is operationally defined as a sequence of successive sucks separated by brief pauses, typically reflecting a rhythmic drinking pattern. For each test stimulus, the number of such bursts is recorded as an integer value. The unit of measure is "number of bursts" (n).
  This outcome is assessed during the first three study visits, where a single test stimulus is administered at each visit. Burst number is not measured during the fourth study visit, in which all three test stimuli are presented simultaneously.
Microstructure of Ingestive Behavior (Burst Duration) | From enrolment to the end of the study participation through three of four study visits within three months.
  Burst duration is defined as the total elapsed time of each individual burst performed by the participant during the ingestion of each of the three test stimuli, as measured using a standardized drinkometer system. A "burst" is operationally defined as a sequence of consecutive sucks separated by brief pauses. For each burst, the duration is measured from the onset of the first suck to the end of the last suck within the burst. The unit of measure is seconds (s).
  This outcome is assessed during the first three study visits, with each visit involving a single test stimulus. Burst duration is not measured during the fourth study visit, in which all three test stimuli are presented simultaneously.
Microstructure of Ingestive Behavior (Burst Energy Intake) | From enrolment to the end of the study participation through three of four study visits within three months.
  Burst energy intake is defined as the total amount of energy intake (in kilocalories) consumed during each individual burst by the participant, measured for each of the three test stimuli using a standardized drinkometer system. A "burst" is operationally defined as a sequence of consecutive sucks separated by brief pauses. For each burst, the energy intake is calculated by multiplying the volume of liquid ingested within the burst by the energy density of the test stimulus. The unit of measure is kilocalories (kcal).
  This outcome is assessed during the first three study visits, each involving a single test stimulus. Burst size is not measured during the fourth study visit, in which all three test stimuli are offered simultaneously.
Microstructure of Ingestive Behavior (Burst Rate) | From enrolment to the end of the study participation through three of four study visits within three months.
  Burst rate is defined as the average rate of energy intake during each individual burst performed by the participant for each of the three test stimuli, as measured using a standardized drinkometer system. For each burst, the total energy intake (in kilocalories) is divided by the duration of the burst (in seconds) to determine the average rate of energy intake for that burst. The unit of measure is kilocalories per second (kcal/s).
  This outcome is assessed during the first three study visits, each involving a single test stimulus. Burst rate is not measured during the fourth study visit, in which all three test stimuli are offered simultaneously.
Microstructure of Ingestive Behavior (Number of Sucks per Burst) | From enrolment to the end of the study participation through three of four study visits within three months.
  Number of sucks per burst is defined as the average count of individual sucks occurring within each burst during the ingestion of each of the three test stimuli, as measured using a standardized drinkometer system. A "burst" is operationally defined as a sequence of consecutive sucks separated by brief pauses. For each burst, the total number of sucks is recorded, and the outcome is typically reported as the mean number of sucks per burst. The unit of measure is "number of sucks per burst" (n).
  This outcome is assessed during the first three study visits, where a single test stimulus is administered at each visit. Number of sucks per burst is not measured during the fourth study visit, in which all three test stimuli are presented simultaneously.
Microstructure of Ingestive Behavior (Inter-Burst Intervals) | From enrolment to the end of the study participation through three of four study visits within three months.
  Inter-burst interval is defined as the elapsed time between the end of one burst and the onset of the subsequent burst during the ingestion of each of the three test stimuli, as measured using a standardized drinkometer system. A "burst" is operationally defined as a sequence of consecutive sucks separated by brief pauses. The inter-burst interval quantifies the temporal spacing between bursts and is recorded in seconds (s).
  This outcome is assessed during the first three study visits, each involving a single test stimulus. Inter-burst intervals are not measured during the fourth study visit, in which all three test stimuli are offered simultaneously.
Microstructure of Ingestive Behavior (Inter-Sucks Intervals) | From enrolment to the end of the study participation through three of four study visits within three months.
  Inter-suck interval is defined as the elapsed time between the end of one suck and the initiation of the subsequent suck during the ingestion of each of the three test stimuli, as measured using a standardized drinkometer system. A "suck" is operationally defined as a discrete negative pressure event corresponding to the drawing in of liquid. The inter-suck interval quantifies the temporal spacing between individual sucks within a burst or throughout the test stimulus consumption, and is recorded in seconds (s).
  This outcome is assessed during the first three study visits, each involving a single test stimulus. Inter-suck intervals are not measured during the fourth study visit, in which all three test stimuli are presented simultaneously.

SECONDARY OUTCOMES:
Plasma GLP-1 Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in GLP-1 concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma GIP Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in GIP concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma Amylin Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in amylin concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma PYY Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in PYY concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma Ghrelin Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in ghrelin concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma Leptin Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in leptin concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma Insulin Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in insulin concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma CCK Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in CCK concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma Glucagon Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in glucagon concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Plasma Serotonin Concentration | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Change in serotonin concentration (pmol/L) from pre-drink to post-drink (immediately and 30 minutes after ingestion), across the three meal types. Unit of measure is picomoles per liter (pmol/L).
Subjective Appetite Sensation: Hunger | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Self-reported hunger rated on a 100-mm visual analogue scale (VAS). Unit of Measure: millimeters (mm).
Subjective Appetite Sensation: Fullness | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Self-reported fullness rated on a 100-mm visual analogue scale (VAS). Unit of Measure: millimeters (mm).
Subjective Appetite Sensation: Desire To Eat | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Self-reported desire to eat rated on a 100-mm visual analogue scale (VAS). Unit of Measure: millimeters (mm).
Subjective Appetite Sensation: Nausea | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Self-reported nausea rated on a 100-mm visual analogue scale (VAS). Unit of Measure: millimeters (mm).
Subjective Appetite Sensation: Abdominal Discomfort | Measured at 3 time points per visit: before the drinkometer test, directly at the end of the drinkometer test, and 30 minutes after the end of the drinkometer test.
  Self-reported abdominal discomfort rated on a 100-mm visual analogue scale (VAS).
  Unit of Measure: millimeters (mm).
Gut Microbiome Composition (Alpha and Beta Diversity) | Up to 14 days after study enrollment (microbiome diversity measured from two stool samples per participant: one in the morning, after afternoon; timing based on participant's natural bowel movement occurrence)
  Microbiome diversity is measured via 16S rRNA sequencing of stool samples collected at two distinct circadian time points: one sample in the morning and one in the late afternoon. The unit of measure is the Shannon index for alpha diversity and the UniFrac distance for beta diversity. While participants are instructed to collect samples at these specific times to capture circadian variation, the exact time of collection is dependent on each participant's individual bowel movement patterns and may vary accordingly.
Gut Microbiome Functional Activity (Metabolite Analysis) | Up to 14 days after study enrollment (microbiome diversity measured from two stool samples per participant: one in the morning, after afternoon; timing based on participant's natural bowel movement occurrence)
  Quantification of microbial metabolites in stool samples. The unit of measure is micromoles per gram stool (µmol/g).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zouhal H, Sellami M, Saeidi A, Slimani M, Abbassi-Daloii A, Khodamoradi A, El Hage R, Hackney AC, Ben Abderrahman A. Effect of physical exercise and training on gastrointestinal hormones in populations with different weight statuses. Nutr Rev. 2019 Jul 1;77(7):455-477. doi: 10.1093/nutrit/nuz005. PMID 31125091
- [Background] Strasser B, Wolters M, Weyh C, Kruger K, Ticinesi A. The Effects of Lifestyle and Diet on Gut Microbiota Composition, Inflammation and Muscle Performance in Our Aging Society. Nutrients. 2021 Jun 15;13(6):2045. doi: 10.3390/nu13062045. PMID 34203776
- [Background] Sondergaard Nielsen M, Rasmussen S, Just Christensen B, Ritz C, le Roux CW, Berg Schmidt J, Sjodin A. Bariatric Surgery Does Not Affect Food Preferences, but Individual Changes in Food Preferences May Predict Weight Loss. Obesity (Silver Spring). 2018 Dec;26(12):1879-1887. doi: 10.1002/oby.22272. Epub 2018 Nov 13. PMID 30421858
- [Background] Serra M, File B, Alceste D, Raguz I, Gero D, Thalheimer A, Widmer J, Ismaeil A, Steinert RE, Spector AC, Bueter M. Burst-pause criterion derivation for drinkometer measurements of ingestive behavior. MethodsX. 2022 May 11;9:101726. doi: 10.1016/j.mex.2022.101726. eCollection 2022. PMID 35620756
- [Background] Quiroga R, Nistal E, Estebanez B, Porras D, Juarez-Fernandez M, Martinez-Florez S, Garcia-Mediavilla MV, de Paz JA, Gonzalez-Gallego J, Sanchez-Campos S, Cuevas MJ. Exercise training modulates the gut microbiota profile and impairs inflammatory signaling pathways in obese children. Exp Mol Med. 2020 Jul;52(7):1048-1061. doi: 10.1038/s12276-020-0459-0. Epub 2020 Jul 6. PMID 32624568
- [Background] Nielsen MS, Christensen BJ, Ritz C, Rasmussen S, Hansen TT, Bredie WLP, le Roux CW, Sjodin A, Schmidt JB. Roux-En-Y Gastric Bypass and Sleeve Gastrectomy Does Not Affect Food Preferences When Assessed by an Ad libitum Buffet Meal. Obes Surg. 2017 Oct;27(10):2599-2605. doi: 10.1007/s11695-017-2678-6. PMID 28411313
- [Background] Moody L, Liang J, Choi PP, Moran TH, Liang NC. Wheel running decreases palatable diet preference in Sprague-Dawley rats. Physiol Behav. 2015 Oct 15;150:53-63. doi: 10.1016/j.physbeh.2015.03.019. Epub 2015 Mar 16. PMID 25791204
- [Background] Monda V, Villano I, Messina A, Valenzano A, Esposito T, Moscatelli F, Viggiano A, Cibelli G, Chieffi S, Monda M, Messina G. Exercise Modifies the Gut Microbiota with Positive Health Effects. Oxid Med Cell Longev. 2017;2017:3831972. doi: 10.1155/2017/3831972. Epub 2017 Mar 5. PMID 28357027
- [Background] Mathes CM, Spector AC. Food selection and taste changes in humans after Roux-en-Y gastric bypass surgery: a direct-measures approach. Physiol Behav. 2012 Nov 5;107(4):476-83. doi: 10.1016/j.physbeh.2012.02.013. Epub 2012 Feb 16. PMID 22366157
- [Background] Mathes CM, Letourneau C, Blonde GD, le Roux CW, Spector AC. Roux-en-Y gastric bypass in rats progressively decreases the proportion of fat calories selected from a palatable cafeteria diet. Am J Physiol Regul Integr Comp Physiol. 2016 May 15;310(10):R952-9. doi: 10.1152/ajpregu.00444.2015. Epub 2016 Feb 10. PMID 26864811
- [Background] Livingstone MBE, Redpath T, Naseer F, Boyd A, Martin M, Finlayson G, Miras AD, Bodnar Z, Kerrigan D, Pournaras DJ, le Roux CW, Spector AC, Price RK. Food Intake Following Gastric Bypass Surgery: Patients Eat Less but Do Not Eat Differently. J Nutr. 2022 Nov;152(11):2319-2332. doi: 10.1093/jn/nxac164. Epub 2022 Jul 23. PMID 36774099
- [Background] Gero D, File B, Justiz J, Steinert RE, Frick L, Spector AC, Bueter M. Drinking microstructure in humans: A proof of concept study of a novel drinkometer in healthy adults. Appetite. 2019 Feb 1;133:47-60. doi: 10.1016/j.appet.2018.08.012. Epub 2018 Sep 1. PMID 30179650
- [Background] Gero D, File B, Alceste D, Frick LD, Serra M, Ismaeil AE, Steinert RE, Spector AC, Bueter M. Microstructural changes in human ingestive behavior after Roux-en-Y gastric bypass during liquid meals. JCI Insight. 2021 Aug 9;6(15):e136842. doi: 10.1172/jci.insight.136842. PMID 34369388
- [Background] Gero D, Bueter M. Post-bariatric changes in ingestive behavior: Shift in macronutrient preferences in rats and dynamic adaptation of the within-meal microstructure in humans. Physiol Behav. 2023 May 1;263:114113. doi: 10.1016/j.physbeh.2023.114113. Epub 2023 Feb 8. PMID 36764423
- [Background] Evero N, Hackett LC, Clark RD, Phelan S, Hagobian TA. Aerobic exercise reduces neuronal responses in food reward brain regions. J Appl Physiol (1985). 2012 May;112(9):1612-9. doi: 10.1152/japplphysiol.01365.2011. Epub 2012 Mar 1. PMID 22383502
- [Background] Dohnalova L, Lundgren P, Carty JRE, Goldstein N, Wenski SL, Nanudorn P, Thiengmag S, Huang KP, Litichevskiy L, Descamps HC, Chellappa K, Glassman A, Kessler S, Kim J, Cox TO, Dmitrieva-Posocco O, Wong AC, Allman EL, Ghosh S, Sharma N, Sengupta K, Cornes B, Dean N, Churchill GA, Khurana TS, Sellmyer MA, FitzGerald GA, Patterson AD, Baur JA, Alhadeff AL, Helfrich EJN, Levy M, Betley JN, Thaiss CA. A microbiome-dependent gut-brain pathway regulates motivation for exercise. Nature. 2022 Dec;612(7941):739-747. doi: 10.1038/s41586-022-05525-z. Epub 2022 Dec 14. PMID 36517598
- [Background] Carter SJ, Hunter GR, Blackston JW, Liu N, Lefkowitz EJ, Van Der Pol WJ, Morrow CD, Paulsen JA, Rogers LQ. Gut microbiota diversity is associated with cardiorespiratory fitness in post-primary treatment breast cancer survivors. Exp Physiol. 2019 Apr;104(4):529-539. doi: 10.1113/EP087404. Epub 2019 Feb 27. PMID 30763983
- [Background] Borer KT, Lin PJ, Wuorinen E. Timing of Meals and Exercise Affects Hormonal Control of Glucoregulation, Insulin Resistance, Substrate Metabolism, and Gastrointestinal Hormones, but Has Little Effect on Appetite in Postmenopausal Women. Nutrients. 2021 Dec 1;13(12):4342. doi: 10.3390/nu13124342. PMID 34959894
- [Background] Beaulieu K, Hopkins M, Gibbons C, Oustric P, Caudwell P, Blundell J, Finlayson G. Exercise Training Reduces Reward for High-Fat Food in Adults with Overweight/Obesity. Med Sci Sports Exerc. 2020 Apr;52(4):900-908. doi: 10.1249/MSS.0000000000002205. PMID 31764466
- [Background] Alceste D, Serra M, Raguz I, Gero D, Thalheimer A, Widmer J, File B, Ismaeil A, Steinert RE, Spector AC, Bueter M. Association between microstructure of ingestive behavior and body weight loss in patients one year after Roux-en-Y gastric bypass. Physiol Behav. 2022 May 1;248:113728. doi: 10.1016/j.physbeh.2022.113728. Epub 2022 Feb 5. PMID 35134394